CLINICAL TRIAL: NCT06924411
Title: Ramped Versus Supine Position for Emergent Endotracheal Intubation in Adult Patients; Prospective, Randomized, Comparative Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Aly Hashem, Resident doctor, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Soh-Med-25-3-04MS
Record Dates: First submitted 2025-04-06; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Intubation Complications
Keywords: Ramped intubation; Non-supine intubation; Semi-setting intubation; Intubation without aspiration; Ramped versus supine intubation; Intubation with less complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine group (Active Comparator): Intubation in supine position
  Interventions: Device: Direct Intubation
- Ramped group (Active Comparator): Intubation in ramped position
  Interventions: Device: Direct Intubation

INTERVENTIONS:
Device: Direct Intubation — Direct laryngoscopy intubation

SUMMARY:
Endotracheal intubation is a life saving procedure for critically unwell and injured patients presenting to the emergency department. Prolonged time to successful intubation and multiple failed attempts are associated with a higher incidence of life-threatening adverse events such as hypoxia and hypotension.

Optimal head and neck positioning and clinical experience are important factors for successful endotracheal intubation in patients especially with a difficult airway. This study aims to investigate the rate of successful endotracheal intubation between ramped and supine positions in patients planned for intubation.

The ramped position, where the bed is kept half-flat and the head is elevated up to 35°, is planned to prove that it improves glottic view and facilitate intubation and ventilation.

Varying bed angles and heights during ramped position intubation may explain conflicting evidence regarding the effect of ramped position on intubation success in acute care settings.

Therefore, it seems that finding a simple alternative method for the classic supine technique that can create conditions like the proposed standard conditions for laryngoscopy would be a suitable solution for intubating patients with higher difficulty.

The patient's anatomy and the technique employed for laryngoscopy have a significant effect on the laryngeal view. The technique itself is influenced by a variety of factors including the laryngoscopic force and the skills, experience, and training of the physicians.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients ≥18 years old and indicated for intubation with variable presentations.

Exclusion Criteria:

* Patients unstable to be positioned in semi setting as spine trauma and polytraumatized patients.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Number of First pass success | 6 months
  Successful intubation from first trial